CLINICAL TRIAL: NCT04260854
Title: Locally Administered Bupivacaine Hydrochloride for Post-operative Pain Control in Cutaneous Surgery: a Randomized Controlled Trial
Brief Title: Bupivacaine Hydrochloride for Pain Control in Cutaneous Surgery
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00211424
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine HCl (Active Comparator): Immediately prior to surgical wound closure, participants randomized to the bupivacaine arm will be injected with bupivacaine HCl along the closure site.
  Interventions: Drug: Bupivacaine Hydrochloride
- Saline (Placebo Comparator): Immediately prior to surgical wound closure, participants randomized to saline, will receive saline injections along the closure site.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Bupivacaine hydrochloride (Hospira, Inc) is an FDA approved, local, injectable indicated for the production of local or regional anesthesia or analgesia for surgery.
  Arms: Bupivacaine HCl
Drug: Saline — Normal saline injections.
  Arms: Saline

SUMMARY:
The purpose of this study is to determine if the addition of bupivacaine HCl injections will improve pain control after skin surgery.

This is a randomized clinical trial. Approximately 100 participants will be randomized to receive either bupivacaine HCl or saline injections to help with the postsurgical pain. Patients will be provided with a take-home journal to complete indicating when and how much pain medication they required for the 3 days immediately following surgery. Participants will return the journal in-person at a follow up visit 7-21 days post-op. This study was a pilot study designed to determine the feasibility of this procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be invited and considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Receiving cutaneous surgery
3. In good general health as assessed by the investigator

Exclusion Criteria:

1. Participants with an allergy to bupivacaine or other amide anesthetics
2. Participants unwilling to sign an IRB approved consent form
3. Participants with a contraindication to narcotic medication
4. Participants who are pregnant or will become pregnant
5. Participants who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reported opioid and non-opioid pain medications taken | 3 Days Post-Surgery
  Patients will report the amount of pain medications taken 3 days immediately following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No